CLINICAL TRIAL: NCT06142071
Title: Mixed Methods Study to Assess Family Members Unmet Needs in an Oncology Setting
Acronym: SALUTE
Status: Active, not recruiting | Type: Observational
Sponsor: Swansea Bay University Health Board (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Other Study IDs: 331660
Record Dates: First submitted 2023-10-26; First posted 2023-11-21 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Telephone questionnaire — Telephone questionnaire, which includes questions on participant's demographics, anxiety/depression scores, what support they find helpful and what additional support they feel would be beneficial

SUMMARY:
The main questions the study aims to answer are:

1. The proportion of family members of cancer patients who say they need more support
2. What support family members feel would be beneficial

Information about patients' cancer diagnosis and treatment will be collected from their medical notes.

Participating family members will be asked to complete a telephone questionnaire. Selected family members may also be asked to participate in an optional follow-up interview.

DETAILED DESCRIPTION:
When someone is diagnosed with cancer, it can be a worrying and stressful time for patients and for their family members. Family members may provide practical and emotional support to patients, and may take on a caregiver role.

Family members may want more information or advice, or may benefit from emotional support themselves. The study aims to identify any gaps in the current support provided to family members so that services can be improved in the future.

Oncology patients in Singleton Hospital, Swansea will be asked by their oncology team to identify one or more family members to participate in the study. If a family member agrees to participate in the study, the research team will call them to complete a telephone questionnaire. The questionnaire should take less than 20 minutes and asks them some general questions (e.g. age, gender) and some questions about how they are feeling, what support services they find helpful and what additional support they feel would be beneficial.

Data regarding participating patients' cancer diagnosis and treatment will be collected from their medical notes.

After the questionnaire data has been analysed, optional follow-up interviews will be conducted with some family members to explore any issues identified in greater detail.

Patients and family members will be recruited during a 6 month recruitment period and all responses will be anonymised.

This is a pilot study which will not change the current support provided to family members, although they may be directed to existing services if appropriate. Patients' treatment will not be changed in any way.

ELIGIBILITY:
Inclusion Criteria for patients

* diagnosed with a solid organ malignancy under the care of the oncology team
* able to identify at least one family member who may be willing to participate in the study

Inclusion Criteria for family members

- a family member of a patient diagnosed with a solid organ malignancy under the care of the oncology team

Exclusion Criteria for patients and family members

* medical or psychiatric condition impairing ability to consent
* the patient's treating oncologist's opinion is that participating in the study would cause severe distress to the patient or their family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients in South West Wales, United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of family members who state they need more support | 6 months after start of study recruitment
  The proportion of family members who state they need more support

SECONDARY OUTCOMES:
The proportion of family members who state they need more support with each of the Carer Support Needs Assessment Tool (CSNAT) domains | 6 months after start of study recruitment
  he proportion of family members who state they need more support with each of the Carer Support Needs Assessment Tool (CSNAT) domains
Types of additional support that family members feel would be beneficial as identified via the telephone questionnaires and interviews | 6 months after start of study recruitment
  This will be determined by qualitative analysis of questionnaire and interview data and may include improved psychological support, online resources, information leaflets etc

CONTACTS AND LOCATIONS:
Overall Officials: Sing Yu Moorcraft, Principal Investigator — Swansea Bay University Health Board
Locations (1):
- South West Wales Cancer Centre, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided